CLINICAL TRIAL: NCT04367012
Title: Prevelance of Non Alcoholic Fatty Liver Disease,Its Complications Among Employees at Banha University Hospital,Egypt
Brief Title: Fatty Liver Among Employees at Banha University
Acronym: fattyliver
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Prof.Reda Mohamed Elbadawy, professor Gastroenterology,Hepatology, Benha University
Other Study IDs: Banha University; Prof.Reda Elbadawy (Other: Hepatology Department)
Record Dates: First submitted 2019-10-10; First posted 2020-04-29 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Fatty Liver Disease; Fatty Infiltration
Keywords: Insulin resistant (IR)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1 NAFLD and group 2 Non NAFLD: study from 20-60 years old.Subjects will be evaluated clinically by abdominal examination for evaluation of fatty liver and grades it into 3 grades .evaluation of fatty pancreas and grade it into 3 grades ,measuring blood pressure and physically by calculating body mass index (BMI) weight/height2
  Interventions: Other: Abdominal Ultrasound
- Group1 NAFLD & Group 2 Non NAFLD: As the study is randomized cross sectional , all subjects whom have fatty liver by abdominal ultrasound included in group 1 NAFLD , and whom do not have fatty liver by abdominal ultrasound included in group 2.both groups was age and sex matched
  Interventions: Other: Abdominal Ultrasound

INTERVENTIONS:
Other: Abdominal Ultrasound — patient in supine position and external carotid artery was examined to meausre the intima using US .Machine GE logic FB inear probe10Mhz.and intimal media thickness mean =10mm
  Other Names: External Carotid Intimal thickness by Dopler

SUMMARY:
This was cross sectional study at Banha University Hospital among employees. Age of the subjects from 20-60 years old both males and females .All investigations done plus abdominal ultrasound for grading of fatty liver and dopler for carotid intima media thickness.

DETAILED DESCRIPTION:
This cross-sectional study was conducted on employees working for the Benha University Hospitals, Qalubeyia Governorate, Egypt. The study population comprised both male and female employees (20 to 60 years old) with no history of viral hepatitis(HBV,HCV) and autoimmune-liver diseases such as primary sclerosing cholangitis and primary billiary cirrhosis . The field work was carried out from September 2018 to March 2019.

This study was approved by the Research Ethics Committee in Benha Faculty of Medicine. An informed consent (in Arabic language) was obtained from all participants. It included all details about the study (title, objectives, methods, expected benefits and risks, and confidentiality of data).

Subjects:

The sample size for the study was calculated according to the following equation 1:

"Sample size" = (〖Z_(1-∝/2)〗^(2 ) P(1-P))/d^2 Where

Z 1-α/2 = standard normal deviate; (at 5% type I error (P<0.05) it is 1.96). P=expected proportion in population based on previous studies 2. d= absolute error or precision (0.05). The total number of the study participants was 165 subjects, who confirm with the inclusion criteria and agreed to participate in the study. These were selected by the systematic random sampling technique.

Data collection tools:

An arranged interview with every study participant was carried out at the Hepatology and Gastrointestinal Department of the Benha University Hospital. All the study participants were exposed to full history taking and clinical examination. Venous blood samples after fasting for 10 hours were collected for complete blood counting, and the assessment of fasting blood glucose, fasting insulin, HOMA-IR test by soecific equation , liver functions testing (ALT,AST ,GGT &Alk.Phosphatase) . kidney functions testing(Serum Urea & Serum Creatinine ) and lipid profile include (serum cholesterol, very low density and high density lipoprotein. Assessment of Liver Fatty Acid Binding Protein (L-FABP), , was carried out using ELIZA. Abdominal Ultrasound for grading of fatty liver from grade 1 to grade 3 according to the comparison with echogencity of right kidney and Doppler on external carotid artery were performed to measure the the intima media thickness.

the different study groups were carried out using the Chi-square test (X2) and the Fisher Exact test (FET) to compare proportions as appropriate. The Student t-test (t) and the Mann-Whitney test (MW) were used to compare two groups of quantitative data regarding parametric and non-parametric data, respectively. While the Kruskal Wallis test and One-Way Analysis Of Variance (ANOVA; F) were used to compare more than two groups, followed by post-hock testing using the Bonferroni method to detect differences in pairs. Spearman correlation coefficient (rho) and Pearson correlation coefficient (r) were used to assess the correlation between the studies parameters as appropriate. the diagnostic performance of L-FAB, HOMA-IR and CIT for NAFLD was examined and the best cut-off and the corresponding Sensitivity, Specificity, Positive Predictive Value (PPV), Negative Predictive Value and Area Under the Curve were estimated. Statistical significance was accepted at P value <0.05 (S).

The statistical analysis was conducted using STATA/SE version 11.2 for Windows (STATA corporation, College Station, Texas).

All the peoples from age 20-60 years old both males and females will be included , apparently healthy either obese or not from banha university employees and students.

They will be evaluated clinically and examined as follow :

* Blood pressure , body mass index(BMI)=heigh/weigh2
* Invesigations as follow , complete blood count(CBC), fasting blood sugar ,glycosyated haemoglobin (HbA1c),Liver function tests including alaninie aminotransferease (ALT) ,aspartateaminotransferase(AST),gamma glutamyl transpeptidase (GGT),alkaline phosphatase ,serum bilirubin, and serum albumin.

lipid profile including (cholesterol,triglycerides,HDL,C and LDL).

* Serum insulin level for calculating insulin resistance (IR) Homostasis Model Assay for Insulin Resistant(HOMA-IR) was assessed using the given mathematical equation; HOMA-IR ¼ fasting insulin (mU/ml) fasting plasma glucose (mmol/l)/22.5 . A HOMA value of 2.18, signifies IR Fatty Acid Binding protein1 (FABP1)
* FABP1 was evaluated after the patient fasting 8 hours by the enzyme-linked immunosorbent assay (ELISA) according to George Haltern ,et al 2010 and the deviation from the normal will be correlated with other investigations and clinical manifestations of the subjects.
* Abdominal Ultrasound was done for grading of fatty liver , to 3 grades from grade 1 to grade3 in comparison to right kidney and diphragm . .
* Carotid Intimal Media Thickenss(CIMT) measured for extracranial portion of Carotid artey by Colour Dopler by measure while the patiet in recumbancy at45 degree and the probe must be in angle less than 90 degree to get the correct results ..

ELIGIBILITY:
Inclusion Criteria:

All subjects was appear healthy with and without DM or hypertension ,also obese or non -

Exclusion Criteria:

Any chronic liver disease , Hepatitis C virus patients (HCV) , Hepatitis B virus patients(HBV) and autoimmune liver disease

-

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Both males and females sex aged from 20-60 years old agree was included in the study after written consent.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-08-25 (Actual)

PRIMARY OUTCOMES:
prevalence of fatty liver among employees at Banha University | 15 month
  Grades of fatty liver was measured as 1,2,3 according to the relation of echogencity beween liver and Right kidney

SECONDARY OUTCOMES:
fatty pancreas among employees at Banha University as compication for fatty liver | 15 months
  Fatty Pancreas was measured by grades 1,2,3 according to the echogencity of retroperitoneal fatt as well as left kidney and liver echogencity

OTHER OUTCOMES:
Atherosclerosis among fatty liver employees at Banha University | 15 month
  Measure the carotid intima media thickness if more than 6mm it will considered atherosclerosis
The associated 7 risk factors | 15 month
  Age>45 years old,DM ,Hypertension ,Urban area,GGT ,ALP and BMI>30kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No
The results of the study